CLINICAL TRIAL: NCT04566835
Title: The Evaluation of Education With Cartoon's Effectiveness on Disease Management of the Children With Asthma
Brief Title: Education With Cartoon's Effectiveness on Disease Management of the Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Aylin Akça Sümengen, Principal Investigator, Faculty Member in Bahcesehir University School of Health Science, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BAU
Record Dates: First submitted 2020-09-16; First posted 2020-09-28 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Asthma in Children
Keywords: pediatric asthma; quality of life in children with asthma; cartoon education in asthma; asthma management education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Assignment to the experimental and control groups was made by a person independent of the researcher. Two balls in different colours, red and white, were placed in a black bag. Assignment to the experimental and control groups was performed by randomly selecting the balls. The following steps:
  Step 0: the first child selected the white ball and was included in the experimental group.
  Step 1: a ball was selected randomly. Step 2: The child was assigned to the experimental group (E) if the ball was white, and to the control group (C) if the ball was red.
  Step 3: A ball in the opposite colour of the selected ball was thrown into the bag (For instance; if the selected ball was red, a white ball was thrown into the bag).
  Step 4: The process was repeated starting from Step 1. The researcher and the subjects did not know which subjects would fall into which group until the intervention was administered. In this way, the possible bias was prevented.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): Taking the Health Promotion Program with cartoons and comics for Children with Asthma
  Interventions: Other: Standart Care given during normal examination; Behavioral: Health Promotion Program with cartoon education for Children with Asthma
- Control Group (Other): Taking standart care
  Interventions: Other: Standart Care given during normal examination

INTERVENTIONS:
Other: Standart Care given during normal examination — This is the standart education given by doctor. The child and his/her parents come to the doctor for normal examination. They take their asthma diagnosis or other information about their condition. and then the doctor explain them about what is asthma, what are the drugs or how should they use them. This is the implementation using for the control group.
Behavioral: Health Promotion Program with cartoon education for Children with Asthma — First of all, the child and their parents take the routine examination as the same as the control group. Then they take the experimental education called Health Promotion Program with cartoon education for Children with Asthma. The children with asthma were educated within the scope of the program in order to demonstrate the effect of the program on asthma management. Children with asthma were educated with the program, which consisted of 4 units, each of 10 minutes, prepared in the light of the literature and with the current guidelines. Each child received the education in a total of 40 minutes. Every unit has its own cartoon video and comic book material. To sum up The Principal Investigator first give the education about asthma management, then makes them watch the Iggy and the Inhalers videos developed for each unit, and does a colouring activity with comic books at the end of each unit.
  Arms: Education Group

SUMMARY:
Objective: The aim of this study is to determine the effect of the education program (HPPCA - Health Promotion Program for Children with Asthma), which was developed by using cartoons and comic based on the health promotion model of Nola J Pender and brain-based learning theories, on disease control and life quality in children aged between 7 and 11, and diagnosed with asthma.

Materials and Methods: The sample of the study consisted of 74 children between the ages of 7 and 11, who presented to a respiratory disease unit of a university hospital in Istanbul. Children were randomly assigned to the experimental (38 children) and control (36 children) groups using the Urn method. It was administered to both groups prior to the intervention. After the HPPCA education administered only to the experimental group, both groups were administered two post-tests as a follow-up in the 1st and 3rd months. Standardized sociodemographic question form, Childhood Asthma Control Test (C-ACT) and Paediatric Asthma Quality of Life Questionnaire (PAQLQ) were used for the follow-up. The data were evaluated using statistical parametric tests.

DETAILED DESCRIPTION:
All guidelines, protocols and recommendations prepared in pediatric asthma emphasize the importance of therapeutic education in asthma management and control. The therapeutic education of children with asthma should be carried out both for skill development and for behavioural changes. Changing the behaviours of individuals is the most difficult part of therapeutic education. Children with asthma should be educated with therapeutic methods and proven nursing models in order to learn disease management and carry out their own asthma control. This model, which targets behavioural changes, has been considered as Pender's Health Promotion Model. The stages of promoting health have been presented clearly; however, the method to be used as a teaching technique in practice has not been clarified. Therefore, it has been suggested in the literature that the model should be used with different training techniques. Looking at the current education and training techniques, the brain-based teaching model, which has been used frequently in educational science in recent years, draws attention. This theory, also known as the neurophysiological theory, was proposed by Donald Olding Hebb in 1951 and developed by Caine & Caine in 1995. With the neurophysiological theory, it has been advocated that the symptom management skills of children with asthma could be made permanent through a good education plan and remindful education methods. The symptoms of asthma are alleviated as the anatomical airway differences disappear when children reach adolescence. They can control asthma better than the young children Therefore, the asthma education is mostly required by the school-age children.

The Health Promotion Model and Brain-Based Training Model in asthma education can best be synthesized with multimedia. The education given with multimedia has been found to be more effective compared to the education given with printed materials. Therefore, the aim of this study is to ensure that the children aged between 7 and 11 learn about disease control and improve their quality of life with an education program (HPPCA - Health Promotion Program for Children with Asthma) developed based on a health promotion model and brain-based learning theories using cartoon and comic book materials.

Trial Design The type of the study is the Randomized Controlled Study, which is one of the quantitative research types. Subjects were assigned to the groups randomly. Pulmonary Function Tests were administered to the children at the beginning of the study, and PFT data were also an outcome. However, when the COVID 19 Pandemic started, current guidelines placed patients with asthma into the risk group and banned PFTs all over the world to prevent the rate of virus spread.

Participants The population of the present study consisted of 653.417 children, which was reported as the total number of children with asthma between 0-18 years in Turkey (who were diagnosed with asthma and prescribed) by Al et al. The study group consisted of 386 children with asthma aged between 7 and 11, who presented to the hospital with asthma according to hospital records after March 2019.

The Place and Time of the Study The pilot study was carried out in the Paediatric Allergy Immunology Outpatient Clinic of a private hospital in Turkey; and the study was carried out in the Paediatric Pulmonology Outpatient Clinic of a state hospital in Turkey. The intervention stages of the study should be carried out in the winter months in terms of the frequency of symptoms of asthma; and the follow-up should be carried out in the spring months, which may increase the atopy and frequency of the symptoms. Therefore, the intervention and follow-up stages of the study were carried out between December 2019 and May 2019.

Interventions Two separate rooms have been prepared for education. An educational environment was created in one of the rooms, and only a test environment was created in the other. The education was implemented in the education room, ensuring that the subjects could not interact with each other. To evaluate the effectiveness of the intervention, a pre-test was applied to both groups prior to the study. In order to evaluate the effectiveness of the education program, both groups were called 1 month later and the first month measurements were performed. Four months after the education, the patients were called again by phone and the measurements were performed in the 4th month. The personal information of the subjects was available only to the researcher. All pre and post intervention tests were recorded with subject numbers. In the study, Health Promotion Program for Children with Asthma (HPPCA) was developed based on the Health Promotion Model and Brain-Based Teaching Method in order to create the most up-to-date and effective method in asthma education. The children with asthma were educated within the scope of the program in order to demonstrate the effect of the program on asthma management. Children with asthma were educated with the program, which consisted of 4 units, each of 10 minutes, prepared in the light of the literature and with the current guidelines. Each child received the education in a total of 40 minutes.

Outcomes The primary outcome of the study was quality of life. Other outcomes are school absenteeism due to asthma, frequency of hospital presentations (unplanned outpatient clinic visits and emergency room visits), quality of life, and asthma control.

Sample Size Power and Sample Size software was used to calculate the sample size. In the study conducted by Kocaslan in 2016, the increase rate created by asthma education on the quality of life variable was taken as reference. In the study by Kocaslan, an 8-point increase was reported in the quality of life as a result of the asthma education, with 95% confidence and 80% power, in 24 experimental and 24 control sizes. Additional subjects were included in the sample, which was calculated at a rate of 20%, in order to prevent the effects of the participants, who discontinued or did not complete the study; and the experimental-control groups were targeted to include 35 individuals. During the course of the study, the first phase of the study was completed as 38 individuals in the experimental group and 36 individuals in the control group. According to the inclusion criteria of the study, the literate children aged between 7 and 11, who were diagnosed with chronic allergic asthma, did not have any communication problems, volunteered to participate in the study, were not in the active attack period (2 weeks are sufficient if there is an attack history), were allergic to substances other than pollen or had no allergies were included in the study after obtaining the informed consent form from their legal guardians.

Randomisation

The random assignment of the subjects to the groups was performed according to the Urn method. This method has been reported to be the most effective method for randomization in small groups. Assignment to the experimental and control groups was made by a person independent of the researcher. According to the Urn method, two balls in different colours, red and white, were placed in a black bag. Assignment to the experimental and control groups was performed by randomly selecting the balls. The following steps were followed during the assignment:

Step 0: the first child selected the white ball and was included in the experimental group.

Step 1: a ball was selected randomly. Step 2: The child was assigned to the experimental group (E) if the ball was white, and to the control group (C) if the ball was red.

Step 3: A ball in the opposite colour of the selected ball was thrown into the bag (For instance; if the selected ball was red, a white ball was thrown into the bag).

Step 4: The process was repeated starting from Step 1. Throwing balls with a contrasting colour to the bag was performed in small groups to minimize the possibility of uneven distribution to the experimental and control groups. The researcher and the subjects did not know which subjects would fall into which group until the intervention was administered. In this way, the possible bias was prevented.

Instruments Sociodemographic Question Form: The questionnaire form, which was developed in line with the literature and intended for children aged 7-11, consisted of 22 questions in total. This form aimed to determine the age, gender, living environment, asthma-related hospital presentations and school absenteeism in the children, who participated in the study. For the validity of the sociodemographic form, a pilot study was conducted with 5 children and these data were not included in the study.

Paediatric Asthma Quality of Life Questionnaire - PAQLQ: It was developed by Juniper at al. in 1996 in Canada, with the aim of assessing the quality of life in children with asthma. The questionnaire aimed to determine the disease-related mental, physical or social disorders of children with asthma, between the ages of 7 and 17. The questionnaire was translated into Turkish by Fidaner et al.; the validity and reliability tests were carried out by Bozkurt. According to the results of their study, Bozkurt and Yıldız, determined the Cronbach's Alpha value of the questionnaire as 0.85 in the first application, and as 0.91 in the second application. The questionnaire inquires the experiences of the children with asthma within the last one week. While administering the questionnaire, the order of the questions should not be changed, and all questions should be answered in order to calculate the score accurately. The questionnaire has three sub-dimensions, which are symptoms, activity limitation and emotional function. The items related to the "Symptoms" sub-dimension are the items 4, 6, 8, 10, 12, 14, 16, 18, 20 and 23. The items 1, 2, 3, 19 and 22 are related to the "Activity Limitation" sub-dimension. Finally, the items 5, 7, 9, 11, 13, 15, 17 and 21 are related to the "Emotional Function" sub-dimension. While applying the questionnaire, the child should be alone. In the questionnaire, the value of each question is between 1 and 7 points, and the score weights of the questions are equal. The lowest score that could be obtained from the scale is 23, and the highest score is 161. The scores of all sub-categories are added together and the mean scores are calculated. Higher score indicates better quality of life.

Childhood Asthma Control Test: This scale was developed by Liu et al. in 2007 in order to measure the asthma control levels of children aged between 4 and 11, in the light of GINA (Global Initiative for Asthma) guidelines. The validity and reliability studies of the Turkish version of the Childhood Asthma Control Test (C-ACT) were carried out by Sekerel et al. in 2012. The scale consists of two parts. The 4 questions asked in the first part are in VAS (visual analogue scale) type and have 4 pictorial options. These questions are asked directly to the child and scored between 0 and 3. The remaining 3 questions are 6-Point Likert-type questions. They are reversely scored, from 5 to 0. This part has to be filled out by the parent. A score between 0 and 27 can be obtained on the scale. The cut-off point for the scale is 19. A score of 19 points or less obtained from the scale indicates that the asthma is not under control of the child. In order to measure the internal consistency of the scale, it was repeated with 5 hospital visits, and a separate Cronbach's alpha value was reported for each visit. For the C-ACT1, C-ACT5, the values were 0.82, 0.83, 0.82, 0.82 and 0.83, respectively. In addition, the test-retest value of the scale was indicated as 0.71.

Cartoon and Comic Materials - Iggy and The Inhalers Cartoons and comics called Iggy and The Inhalers, which were the educational materials to be used in this study, were designed and published by Thomas and Ashwal in 2014 for children aged between 7 and 12. The materials were developed by a paediatric allergist, a healthcare communications specialist, a paediatric asthma nurse and a graphic designer in the light of the international guidelines (National Asthma Education and Prevention Program (NAEPP), Global Initiative for Asthma (GINA)). Iggy and The Inhalers was developed for school children to understand the pathophysiology, symptoms, medications, and inhaler techniques of asthma according to the characteristics of their age. It also teaches the triggers that worsen the symptoms as well as the methods to avoid these triggers. The translation for the Turkish language was simultaneously checked by 10 experts, who knew both languages well, and the dubbing process was performed by the researcher in a professional studio. The recordings were sent to the Booster Shot Media company to be embedded in the video. In addition, the graphic design of the cartoons was rearranged, and the English words used in the cartoons were translated into Turkish. Cartoons and comics called Iggy and The Inhalers were used for the first time in Turkey. The effectiveness and experiments of these materials were made by Thomas and Ashwall in 2014, and were used again by Catherine et al in 2017.

Statistical Methods The data obtained in the study were evaluated by statistical analysis methods. SPSS 26.0 analysis program was used for this evaluation. Descriptive statistical methods were used to analyse the sociodemographic characteristics of the subjects. In order to evaluate the effectiveness of the intervention in the study data, the differences between before and after the intervention were evaluated through the parametric tests according to the normal distribution characteristics of the data. Among the parametric tests, the t-test, ANOVA and Chi-square tests were used. Independent sample t-test and repeated measures ANOVA were used to determine the relationship between the asthma control and quality of life variables.

Resources of Support and Approval of the Ethics Committee No financial support was received for the preparation of the work. Ethics committee approval was obtained from Koç University Clinical Research Ethics Committee, with the code number 2019.329.IRB1.056. Institutional permission was obtained from Health Sciences University Hamidiye Etfal Training and Research Hospital. A contract was signed with Booster Shot Media for using and translating Iggy and The Inhalers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic allergic asthma,
* Did not have any communication problems,
* Volunteered to participate in the study,
* Were not in the active attack period (2 weeks are sufficient if there is an attack history),
* Were allergic to substances other than pollen or had no allergies
* Were included in the study after obtaining the informed consent form from their legal guardians.

Exclusion Criteria:

- Opposite of the inclusion criteria

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2019-12-21 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Paediatric Asthma Quality of Life Questionnaire - PAQLQ | Pre Test
  The questionnaire has three sub-dimensions, which are symptoms, activity limitation and emotional function. The items related to the "Symptoms" sub-dimension are the items 4, 6, 8, 10, 12, 14, 16, 18, 20 and 23. The items 1, 2, 3, 19 and 22 are related to the "Activity Limitation" sub-dimension. Finally, the items 5, 7, 9, 11, 13, 15, 17 and 21 are related to the "Emotional Function" sub-dimension. While applying the questionnaire, the child should be alone. In the questionnaire, the value of each question is between 1 and 7 points, and the score weights of the questions are equal. The lowest score that could be obtained from the scale is 23, and the highest score is 161. The scores of all sub-categories are added together and the mean scores are calculated. Higher score indicates better quality of life
Childhood Asthma Control Test | Pre Test
  The scale consists of two parts. The 4 questions asked in the first part are in VAS (visual analogue scale) type, and have 4 pictorial options. These questions are asked directly to the child and scored between 0 and 3. The remaining 3 questions are 6-Point Likert-type questions. They are reversely scored, from 5 to 0. This part has to be filled out by the parent. A score between 0 and 27 can be obtained on the scale. The cut-off point for the scale is 19. A score of 19 points or less obtained from the scale indicates that the asthma is not under control of the child.
Childhood Asthma Control Test-Change from Pre Test on first month | 1st month
  The scale consists of two parts. The 4 questions asked in the first part are in VAS (visual analogue scale) type, and have 4 pictorial options. These questions are asked directly to the child and scored between 0 and 3. The remaining 3 questions are 6-Point Likert-type questions. They are reversely scored, from 5 to 0. This part has to be filled out by the parent. A score between 0 and 27 can be obtained on the scale. The cut-off point for the scale is 19. A score of 19 points or less obtained from the scale indicates that the asthma is not under control of the child.
Pediatric Asthma Quality of Life Questionnaire - Change from Pre Test on first month | 1st month
  The questionnaire has three sub-dimensions, which are symptoms, activity limitation and emotional function. The items related to the "Symptoms" sub-dimension are the items 4, 6, 8, 10, 12, 14, 16, 18, 20 and 23. The items 1, 2, 3, 19 and 22 are related to the "Activity Limitation" sub-dimension. Finally, the items 5, 7, 9, 11, 13, 15, 17 and 21 are related to the "Emotional Function" sub-dimension. While applying the questionnaire, the child should be alone. In the questionnaire, the value of each question is between 1 and 7 points, and the score weights of the questions are equal. The lowest score that could be obtained from the scale is 23, and the highest score is 161. The scores of all sub-categories are added together and the mean scores are calculated. Higher score indicates better quality of life
Childhood Asthma Control Test-Change from pretest, first month and fourth month | 4th month
  The scale consists of two parts. The 4 questions asked in the first part are in VAS (visual analogue scale) type, and have 4 pictorial options. These questions are asked directly to the child and scored between 0 and 3. The remaining 3 questions are 6-Point Likert-type questions. They are reversely scored, from 5 to 0. This part has to be filled out by the parent. A score between 0 and 27 can be obtained on the scale. The cut-off point for the scale is 19. A score of 19 points or less obtained from the scale indicates that the asthma is not under control of the child.
Pediatric Asthma Quality of Life Questionnaire - Change from pretest, first month and fourth month | 4th month
  The questionnaire has three sub-dimensions, which are symptoms, activity limitation and emotional function. The items related to the "Symptoms" sub-dimension are the items 4, 6, 8, 10, 12, 14, 16, 18, 20 and 23. The items 1, 2, 3, 19 and 22 are related to the "Activity Limitation" sub-dimension. Finally, the items 5, 7, 9, 11, 13, 15, 17 and 21 are related to the "Emotional Function" sub-dimension. While applying the questionnaire, the child should be alone. In the questionnaire, the value of each question is between 1 and 7 points, and the score weights of the questions are equal. The lowest score that could be obtained from the scale is 23, and the highest score is 161. The scores of all sub-categories are added together and the mean scores are calculated. Higher score indicates better quality of life

SECONDARY OUTCOMES:
Number of School absenteeism | Pre Test
  If child don't go to the school because of the asthma attack. The investigators evaluate it with a question. The investigators' question was; Have participants ever been absent from school due to asthma in the last four weeks' And the child answer it yes or no
Number of Hospital Visits | Pre Test
  unplanned outpatient clinic visits and emergency room visits. The investigators ask a question to parents; Have participants applied for an unplanned hospital admission due to asthma in the last four weeks?
Number of School absenteeism -Change from Pre Test on first month | 1st month
  If child don't go to the school because of the asthma attack. And the investigators evaluate the change for school absenteeism with new question; Have participants ever been absent from school due to asthma in the last eight weeks. And this is a yes or no question.
Number of Hospital Visits -Change from Pre Test on first month | 1st month
  unplanned outpatient clinic visits and emergency room visits.Have participants applied for an unplanned hospital admission due to asthma in the eight weeks? They should answer it yes or no.
Number of School absenteeism -Change from pretest to first month and fourth month | 4th month
  If child don't go to the school because of the asthma attack. The investigators ask the question again; Have participants been absent from school due to asthma in the last four months? And the child should answer it yes or no.
Number of Hospital Visits-Change from pretest, first month and fourth month | 4th month
  unplanned outpatient clinic visits and emergency room visits. The investigators ask them a question; Have participants applied for an unplanned hospital admission due to asthma in the last four months? The investigators expect them to answer it yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse F Ocakci, Professor, Study Director — Advisor
Locations (1):
- Koc University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators took an informed consent form from parents and declared that never share any personal information about the participants.

REFERENCES:
- [Background] Abadoğlu, Ö., Başyiğit, İ., Bavbek, S., Bayındır, Ü., Bayram, H., Bingöl, G., . . . Yüksel, H. (2016). Türk Toraks Derneğİ Astim Tani ve Tedavİ Rehberİ. Official Journal of the Turkish Thoracic Society(17).
- [Background] Akdeniz, E., & Öncel, S. (2019). Türkiye'de Hemşirelik Alanında Astımlı Çocuklarla İlgili Yapılan Lisansüstü Tezlerin İncelenmesi. Turkiye Klinikleri Hemsirelik Bilimleri, 11(2).
- [Background] Aktan, Z. D., Berk, H., Erdoğan, F., & Öktem, S. (2019). Relationship Between Serum IgE Level and Anxiety, Depression, Somatization and Quality of Life in Pediatric Asthma. Current Approaches in Psychiatry/Psikiyatride Guncel Yaklasimlar, 11.
- [Background] Al, S., & Özcebe, H. (2017). Sosyal Güvenlik Kurumu Kayıtlarında 0-18 Yaş Aralığı İçin Astım Hastalığının Analizi. Sosyal Güvence Dergisi, 6(12), 32.
- [Background] Alkan, H. Ö. (2016). Hasta Eğitimi ve Davranış Değişikliği Geliştirme. Journal of Cardiovascular Nursing, 7(Sup 2), 41-47.
- [Background] Bozkurt, G., & Yıldız, S. (2004). Astımlı Okul Çocuklarına Hastalığın Yönetimi Konusunda Verilen Eğitimin Yaşam Kalitelerine Etkisi. İstanbul Üniversitesi F.N.H.Y.O. Dergisi, 13(53), 101-113.
- [Background] Çoruhlu, T. Ş., Nas, S. E., & Keleş, E. J. A. Ü. E. F. D. (2016). Beyin Temelli Öğrenme Yaklaşımına Dayalı Web Destekli Öğretim Materyalinin Etkililiğinin Değerlendirilmesi: Işık ve Ses Ünitesi. 5(1), 104-132.
- [Background] Çövener, Ç. (2012). Tip 1 Diyabet Yönetiminde Sağlığı Geliştirme Modeli ve Tam öğrenme Kuramına Dayalı Eğitimin Etkisi. (Doctoral Doctoral). Marmara University, Istanbul.
- [Background] Demirbaş, B. C., Çekiç, Ş., Canıtez, Y., & Sapan, N. (2017). Okul çağındaki astımlı olguların çocukluk çağı astım kontrol testi ile değerlendirilmesi. Güncel Pediatri, 15(3), 11-16.
- [Background] Hockenberry, M. J., & Wilson, D. (2018). Wong's nursing care of infants and children-E-book: Elsevier Health Sciences.
- [Background] Hsu, J., Sicrar, K., Herman, E., & Garbe, P. (2018). EXHALE: A Technical Package to Control Asthma
- [Background] Kanık, E. A., Taşdelen, B., & Erdoğan, S. (2011). Klinik denemelerde randomizasyon.
- [Background] Karadağ, A., Çalışkan, N., & Baykara, Z. G. (2017). Hemşirelik Teorileri ve Modelleri (Vol. Baskı 1). İstanbul: Akademi Basın ve Yayıncılık
- [Background] Tan NC, Chen Z, Soo WF, Ngoh AS, Tai BC. Effects of a written asthma action plan on caregivers' management of children with asthma: a cross-sectional questionnaire survey. Prim Care Respir J. 2013 Jun;22(2):188-94. doi: 10.4104/pcrj.2013.00040. PMID 23616054
- [Result] Abdelsalam, S. (2017). Outcome of Self-Management Training On Quality Of Life And Self-Efficacy In Patients With Bronchial Asthma. 6.
- [Result] Beller EM, Gebski V, Keech AC. Randomisation in clinical trials. Med J Aust. 2002 Nov 18;177(10):565-7. doi: 10.5694/j.1326-5377.2002.tb04955.x. No abstract available. PMID 12429008
- [Result] Brown S, Lehr VT, French N, Giuliano CA. Can a Short Video Improve Inhaler Use in Urban Youth? J Pediatr Pharmacol Ther. 2017 Jul-Aug;22(4):293-299. doi: 10.5863/1551-6776-22.4.293. PMID 28943825
- [Result] Butz A, Pham L, Lewis L, Lewis C, Hill K, Walker J, Winkelstein M. Rural children with asthma: impact of a parent and child asthma education program. J Asthma. 2005 Dec;42(10):813-21. doi: 10.1080/02770900500369850. PMID 16393717
- [Result] Cicutto L, To T, Murphy S. A randomized controlled trial of a public health nurse-delivered asthma program to elementary schools. J Sch Health. 2013 Dec;83(12):876-84. doi: 10.1111/josh.12106. PMID 24261522
- [Result] Çinar, S. (2015). Effect of educational on symptom control and quality of life on asthmatic patients
- [Result] Clark NM, Shah S, Dodge JA, Thomas LJ, Andridge RR, Little RJ. An evaluation of asthma interventions for preteen students. J Sch Health. 2010 Feb;80(2):80-7. doi: 10.1111/j.1746-1561.2009.00469.x. PMID 20236406
- [Result] George, D., & Mallery, M. (2010). SPSS for Windows Step BysStep: A Simple Guide and Reference
- [Result] Gerald LB, McClure LA, Mangan JM, Harrington KF, Gibson L, Erwin S, Atchison J, Grad R. Increasing adherence to inhaled steroid therapy among schoolchildren: randomized, controlled trial of school-based supervised asthma therapy. Pediatrics. 2009 Feb;123(2):466-74. doi: 10.1542/peds.2008-0499. PMID 19171611
- [Result] Gulla KM, Kabra SK. Peak Expiratory Flow Rate as a Monitoring Tool in Asthma. Indian J Pediatr. 2017 Aug;84(8):573-574. doi: 10.1007/s12098-017-2398-x. Epub 2017 Jun 14. No abstract available. PMID 28612223
- [Result] Jaudes, P. K., Bilaver, L. A., & Champagne, V. (2015). Do children in foster care receive appropriate treatment for asthma? Children and Youth Services Review, 52, 103-109. doi:https://doi.org/10.1016/j.childyouth.2015.03.004
- [Result] Julian V, Amat F, Petit I, Pereira B, Fauquert JL, Heraud MC, Labbe G, Labbe A. Impact of a short early therapeutic education program on the quality of life of asthmatic children and their families. Pediatr Pulmonol. 2015 Mar;50(3):213-221. doi: 10.1002/ppul.23013. Epub 2014 Feb 24. PMID 24574193
- [Result] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in children with asthma. Qual Life Res. 1996 Feb;5(1):35-46. doi: 10.1007/BF00435967. PMID 8901365
- [Result] King TL, Kho EK, Tiong YH, Julaihi SN. Comparison of effectiveness and time-efficiency between multimedia and conventional counselling on metered-dose inhaler technique education. Singapore Med J. 2015 Feb;56(2):103-8. doi: 10.11622/smedj.2015024. PMID 25715856
- [Result] Kocaaslan, E. N. (2016a). Astımlı çocuklarda hastalık yönetimi konusunda verilen eğitimin çocukların yaşam kalitesi ve öz etkililik düzeylerkine etkisi. Trakya Üniversitesi Sağlık Bilimleri Enstitüsü
- [Result] Li Z, Leite WL, Thompson LA, Gross HE, Shenkman EA, Reeve BB, DeWalt DA, Huang IC. Determinants of longitudinal health-related quality-of-life change in children with asthma from low-income families: a report from the PROMIS(R) Pediatric Asthma Study. Clin Exp Allergy. 2017 Mar;47(3):383-394. doi: 10.1111/cea.12827. Epub 2016 Oct 21. PMID 27664979
- [Result] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Result] Liu PC, Kieckhefer GM, Gau BS. A systematic review of the association between obesity and asthma in children. J Adv Nurs. 2013 Jul;69(7):1446-65. doi: 10.1111/jan.12129. Epub 2013 Apr 8. PMID 23560878
- [Result] McClure N, Seibert M, Johnson T, Kannenberg L, Brown T, Lutenbacher M. Improving Asthma Management in the Elementary School Setting: An Education and Self-management Pilot Project. J Pediatr Nurs. 2018 Sep-Oct;42:16-20. doi: 10.1016/j.pedn.2018.06.001. Epub 2018 Jun 12. PMID 30219294
- [Result] McGhan SL, Wong E, Sharpe HM, Hessel PA, Mandhane P, Boechler VL, Majaesic C, Befus AD. A children's asthma education program: Roaring Adventures of Puff (RAP), improves quality of life. Can Respir J. 2010 Mar-Apr;17(2):67-73. doi: 10.1155/2010/327650. PMID 20422062
- [Result] Mickel CF, Shanovich KK, Evans MD, Jackson DJ. Evaluation of a School-Based Asthma Education Protocol. J Sch Nurs. 2017 Jun;33(3):189-197. doi: 10.1177/1059840516659912. Epub 2016 Jul 22. PMID 27450449
- [Result] Korta Murua J, Valverde Molina J, Praena Crespo M, Figuerola Mulet J, Rodriguez Fernandez-Oliva CR, Rueda Esteban S, Neira Rodriguez A, Vazquez Cordero C, Martinez Gomez M, Roman Pinana JM. [Therapeutic education in asthma management]. An Pediatr (Barc). 2007 May;66(5):496-517. doi: 10.1157/13102515. Spanish. PMID 17517205
- [Result] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Result] Ochoa Sangrador C, Vazquez Blanco A. Day-care center attendance and risk of Asthma-A systematic review. Allergol Immunopathol (Madr). 2018 Nov-Dec;46(6):578-584. doi: 10.1016/j.aller.2018.03.006. Epub 2018 Jul 7. PMID 30318106
- [Result] Rosenberger, W. F., & Lachin, J. M. (2015). Randomization in clinical trials: theory and practice: John Wiley & Sons
- [Result] Saleh ASEM. School asthma intervention programme effectively improved children's knowledge and attitudes, and led to decreased hospital admission, length of stay and school absences. Evid Based Nurs. 2020 Jul;23(3):92. doi: 10.1136/ebnurs-2019-103092. Epub 2019 Aug 19. No abstract available. PMID 31427502
- [Result] Sekerel BE, Soyer OU, Keskin O, Uzuner N, Yazicioglu M, Kilic M, Artac H, Ozmen S, Can D, Zeyrek D, Cokugras H, Canitez Y, Aydogan M, Kuyucu S, Inal A, Gurkan F, Orhan F, Yilmaz O, Boz AB, Tahan F, Cevit O. The reliability and validity of Turkish version of Childhood Asthma Control Test. Qual Life Res. 2012 May;21(4):685-90. doi: 10.1007/s11136-011-9970-z. Epub 2011 Jul 27. PMID 21792732
- [Result] Somashekar AR, Ramakrishnan KG. Evaluation of Asthma Control in Children Using Childhood- Asthma Control Test (C-ACT) and Asthma Therapy Assessment Questionnaire (ATAQ). Indian Pediatr. 2017 Sep 15;54(9):746-748. doi: 10.1007/s13312-017-1167-2. PMID 28984253
- [Result] Szefler SJ, Cloutier MM, Villarreal M, Hollenbach JP, Gleason M, Haas-Howard C, Vinick C, Calatroni A, Cicutto L, White M, Williams S, McGinn M, Langton C, Shocks D, Mitchell H, Stempel DA. Building Bridges for Asthma Care: Reducing school absence for inner-city children with health disparities. J Allergy Clin Immunol. 2019 Feb;143(2):746-754.e2. doi: 10.1016/j.jaci.2018.05.041. Epub 2018 Jul 25. PMID 30055181
- [Result] Tabachnick, B., Fidell, L., Tabachnick, B., & Fidell, L. (2014). Using multivariate statistics (6th New International ed.). Essex: Pearson, 235, 284.
- [Result] Walter H, Sadeque-Iqbal F, Ulysse R, Castillo D, Fitzpatrick A, Singleton J. Effectiveness of school-based family asthma educational programs in quality of life and asthma exacerbations in asthmatic children aged five to 18: a systematic review. JBI Database System Rev Implement Rep. 2016 Nov;14(11):113-138. doi: 10.11124/JBISRIR-2016-003181. PMID 27941517
- See also: AİD. (2020). COVID-19 Asthma Management During COVİD 19 Pandemic — https://www.aid.org.tr/covid-19-pandemisinde-agir-astim-yonetimi/
- See also: Asthma Statistics (2018) — https://asthma.org.au/about-asthma/understanding-asthma/statistics/
- See also: World Asthma Day Report — https://artvindh.saglik.gov.tr/TR,165354/dunya-astim-gunu-basin-bildirisi-2019.html
- See also: Centers for Disease Control and Prevention Vital Signs — https://www.cdc.gov/vitalsigns/index.html
- See also: Gibson, J. (2019). European Lung White Book Burden Lung Diease. Childhood Asthma — https://www.erswhitebook.org/files/public/Chapters/11_childhood_asthma.pdf
- See also: GINA. (2018). Global Initiative for Asthma 2018 GINA Report, Global Strategy for Asthma Management and Prevention. — https://ginasthma.org/2018-gina-report-global-strategy-for-asthma-management-and-prevention/
- See also: GINA. (2019). Global Initiative for Asthma 2018 GINA Report, Global Strategy for Asthma Management and Prevention — https://ginasthma.org/wp-content/uploads/2019/04/GINA-2019-main-Pocket-Guide-wms.pdf
- See also: GINA. (2020a). COVID-19: GINA Answers to Frequently Asked Questions on asthma Management — https://ginasthma.org/covid-19-gina-answers-to-frequently-asked-questions-on-asthma-management/final-covid-19-answers-to-frequent-questions-25-3-2020-1/
- See also: GINA. (2020b). COVID-19: GINA Answers to Frequently Asked Questions on Asthma Management. — https://ginasthma.org/wp-content/uploads/2020/03/Final-COVID-19-answers-to-frequent-questions-25.3.2020-1.pdf
- See also: enkinson, C. (2019). Quality of life — https://www.britannica.com/topic/quality-of-life
- See also: SPSS, I. (2019). IBM SPSS Statistics 26 (Version 26): IBM Developer. — https://www.ibm.com/tr-tr/products/spss-statistics/details
- See also: Thomas, A., & Ashwall, G. (2014). Iggy and the inhalers: Multimedia Asthma Education Program — https://iggyandtheinhalers.com/